CLINICAL TRIAL: NCT00372853
Title: A Phase 1 Dose Escalation Trial To Evaluate The Safety And Tolerability Of CP-675,206 Administered In Combination With SU011248 To Patients With Metastatic Renal Cell Carcinoma
Brief Title: Dose-Finding Study Of CP-675,206 And SU011248 In Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671025
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tremelimumab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: CP-675,206; Drug: SU011248
- Arm B (Experimental)
  Interventions: Drug: CP-675,206; Drug: SU011248

INTERVENTIONS:
Drug: CP-675,206 — CP-675,206 administered intravenously every 3 months. Escalating doses from 6mg/kg to 15mg/kg will be tested.
  Arms: Arm A
Drug: SU011248 — SU011248 administered at a dose of 37.5mg/day every day.
  Arms: Arm A
Drug: CP-675,206 — CP-675,206 administered intravenously every 3 months. Escalating doses from 6mg/kg to 15mg/kg will be tested.
  Arms: Arm B
Drug: SU011248 — SU011248 administered at a dose of 50mg/day for 4 weeks followed by 2 weeks off, repeated every 6 weeks.
  Arms: Arm B

SUMMARY:
This study will determine the highest tolerable dose of CP-675,206 when given in combination with SU011248.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma with metastases
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1

Exclusion Criteria:

* Prior treatment with more than one systemic therapy for metastatic renal cell carcinoma
* History of or known brain metastases, spinal cord compression or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening Computed Axial Tomography (CT) or Magnetic Resonance Imaging (MRI) scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the highest tolerable dose of CP-675,206 that can be combined with SU011248. The safety observation period will be 6 weeks from the first dose of study drug | 6 weeks after first dose

SECONDARY OUTCOMES:
To allow for the possibility of genotyping should an unexpected outcome or an increase in unexplained adverse events be reported | 18 months
To evaluate the pharmacokinetics (PK) of CP-675,206 and SU011248 when given in combination | up to 18 months
To monitor for an antibody response to CP-675,206 | up to 18 months
To assess any preliminary evidence of anti-tumor activity: 6-18 months after last subject enrolled | 6-18 months after last subject enrolled

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Scottsdale, Arizona
  - Research Site, New Brunswick, New Jersey
  - Research Site, Cleveland, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee